CLINICAL TRIAL: NCT07083518
Title: Efficacy and Mechanisms of Transcranial Direct Current Stimulation (tDCS) on Cancer-Related Cognitive Impairment(CRCI) in Breast Cancer Survivors: A Randomized Controlled Trial
Brief Title: Transcranial Direct Current Stimulation for Cancer-related Cognitive Impairment in Breast Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AHMU-tDCS-BC
Record Dates: First submitted 2025-06-24; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Transcranial Direct Current Stimulation (tDCS); Breast Cancer Survivor; Cognitive Impairment
Keywords: tDCS; breast cancer; cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction; Breast Neoplasms | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anodal tDCS (Active Comparator): Participants will receive active tDCS for 20 minutes daily, 5 sessions per week, over 4 consecutive weeks (total 20 sessions). The anodal electrode was placed on the DLPFC (F3) surrounded by four cathodes with 1-cm diameter (FCz, AFz, F7, and C5). The stimulation direct current magnitude was set at 2 mA with a 30-s immediate decline at the beginning and end of each phase.
  Interventions: Device: Anodal transcranial direct current stimulation
- sham stimulation (Sham Comparator): Participants will receive sham stimulation for 20 minutes daily, 5 sessions per week, over 4 consecutive weeks (total 20 sessions). In the sham condition, a 30-s rising current until 2 mA is reached, with a 30-s decline immediately at the beginning and end of the stimulation section.
  Interventions: Device: Sham transcranial direct current stimulation

INTERVENTIONS:
Device: Anodal transcranial direct current stimulation — tDCS is described as a non-invasive form of brain stimulation that uses a low-intensity, direct current applied directly to the head through scalp electrodes.
  Arms: Anodal tDCS
Device: Sham transcranial direct current stimulation — Sham tDCS was delivered using the same protocol and current intensity, but the period of active stimulation was only during the ramp-up and ramp-down periods of 30 and 30 seconds.
  Arms: sham stimulation

SUMMARY:
This study aims to evaluate the efficacy of transcranial direct current stimulation (tDCS) in improving cancer-related cognitive impairment (CRCI) in breast cancer survivors. Participants will be randomly assigned to receive active or sham stimulation over the prefrontal cortex. Cognitive outcomes will be assessed using standardized neuropsychological tests and self-reported measures. Functional magnetic resonance imaging (fMRI) and electroencephalography (EEG) will be used to explore neural correlates of intervention effects.

DETAILED DESCRIPTION:
This study is designed to evaluate the therapeutic effects of transcranial direct current stimulation (tDCS) on cancer-related cognitive impairment (CRCI) in breast cancer survivors. CRCI is a common and persistent complication among patients treated with systemic cancer therapies and has a substantial impact on quality of life, even after completion of treatment. Participants will be female breast cancer survivors who have completed primary treatments and report cognitive complaints. Eligible individuals will be randomized in a 1:1 ratio to receive either active or sham tDCS. The stimulation will be applied over the left dorsolateral prefrontal cortex (DLPFC), a brain region involved in executive function, memory, and attention. Each participant will receive multiple sessions of tDCS across a defined intervention period. The primary outcome will be the change in perceived cognitive function, measured by the total score of the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) questionnaire. Secondary outcomes will include objective performance on neuropsychological tests (Trail Making Test, Auditory Verbal Learning Test, Digit Span Test), as well as patient-reported fatigue (Piper Fatigue Scale) and emotional symptoms (HAMD, HAMA). Neuroimaging (fMRI) and electrophysiological (EEG) data will also be collected in a subset of participants to explore neural correlates of treatment effects.

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer survivors aged 18-65 years.
2. Initially diagnosed with stage I-III non-metastatic breast cancer.
3. Between 6 months and 5 years after completion of initial curative surgery +/- radiation/chemotherapy.
4. allowed to be on endocrine therapy and/or anti-HER2 targeted therapy.
5. Self-reported cognitive complaints following cancer treatment.
6. Right-handedness (for standardized tDCS targeting)
7. Education level ≥ 6 years
8. Able and willing to undergo all study procedures (neuropsychological testing, MRI, EEG, etc.) and to provide written informed consent

Exclusion Criteria:

1. Contraindications to MRI or EEG (e.g., pacemaker, metallic implants, claustrophobia).
2. Active neurological/psychiatric disorders (e.g., major depressive disorder, bipolar disorder, schizophrenia, Parkinson's disease, post-stroke sequelae)
3. Concurrent use of cognition-enhancing medications (e.g., donepezil, memantine)
4. Severe somatic diseases (cardiac/hepatic/renal insufficiency)
5. Pregnant or breastfeeding
6. Concurrent participation in another interventional clinical trial

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  FACT-Cog is a validated self-report instrument designed to assess perceived cognitive function in cancer patients and survivors. It evaluates the individual's subjective experience of cognitive abilities during and after cancer treatment. Higher total scores reflect better perceived cognitive functioning. Only the overall score will be used as the outcome measure in this study.

SECONDARY OUTCOMES:
Trail Making Test | baseline, immediately post-intervention, 1-month post-intervention, 3-months post-intervention
  Executive function will be assessed using the Trail Making Test, including Part A (visual attention and processing speed) and Part B (task switching and cognitive flexibility). Higher completion times reflect poorer performance. The difference in completion time from baseline will be used as the outcome.
Digit Span Test | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  Working memory will be assessed using the Digit Span Test (forward and backward conditions). Scores reflect the maximum number of digits recalled in correct order.
Auditory Verbal Learning Test | baseline, immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  Verbal memory will be assessed using the Auditory Verbal Learning Test (AVLT), including immediate recall (sum of trials), delayed recall, and recognition accuracy. Scores reflect the number of correctly recalled or recognized items.
Piper Cancer-Related Fatigue Scale Score (PFS) | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  The Piper Cancer-Related Fatigue Scale (PFS) is a validated self-report instrument used to assess the severity of cancer-related fatigue. It contains 22 items scored on a 0-10 scale, with higher total scores indicating greater fatigue severity. Only the total score will be used as the outcome measure.
Hamilton Depression Rating Scale (HAMD) | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  The changes in HAMD will constitute the secondary research outcome. The Hamilton Depression Scale (HAMD), compiled by Hamilton in 1960, is the most common clinical scale to assess depression. In this study, 17 versions were selected, and there were 17 questions. Each question scored between 0 and 4 points. Higher scores indicate more depressive symptoms. The severity of the disease and the therapeutic effect can be evaluated after treatment.
  Endpoint: Difference between each time point's total score and baseline; negative Δ indicates symptom relief.
  Analysis: Repeated measures mixed-effects model, exploring the moderating effect of mood on cognitive outcomes.
Hamilton Anxiety Scale(HAMA) | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  The Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959. It was one of the most commonly used scales in psychiatric clinics, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder.
  Endpoint: Difference between each time point's total score and baseline; negative Δ indicates symptom relief.
  Analysis: Repeated measures mixed-effects model, exploring the moderating effect of mood on cognitive outcomes.
The Changes of Functional Magnetic Resonance Imaging (fMRI) | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  The change of resting-state functional connectivity strength between the stimulated target and the whole brain areas will be measured by functional magnetic resonance imaging (fMRI): within-subject changes in (1) resting-state functional connectivity among key networks, (2) regional brain volumes (e.g., prefrontal cortex, hippocampus), and (3) white matter integrity (fractional anisotropy, mean diffusivity), reflecting tDCS effects on brain structure and function.
The change of resting-state electroencephalography (EEG) | baseline (pre-intervention), immediately post-intervention, 1-month post-intervention, and 3-months post-intervention
  The change of resting-state functional connectivity strength between the stimulated target and the whole brain areas will be measured by resting-state electroencephalography (EEG): preprocessing (filtering, artifact removal), computation of relative power in δ/θ/α/β/γ bands, and extraction of P300 amplitude and latency. Endpoint: Difference in spectral power and ERP metrics relative to baseline. Analysis: Repeated measures ANOVA with post-hoc Bonferroni correction.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China